CLINICAL TRIAL: NCT04482868
Title: Percutaneous Screw Fixation for Acute Scaphoid Fractures Through K-wire-assisted Reduction and Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Chunjie Liu, Chief physician, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-09-03
Record Dates: First submitted 2020-07-19; First posted 2020-07-23 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Hand; Wrist; Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries | interventions — Maintenance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open reduction group (Placebo Comparator)
  Interventions: Procedure: Percutaneous screw fixation through K-wire-assisted reduction and maintenance
- percutaneous group (Experimental)
  Interventions: Procedure: Percutaneous screw fixation through K-wire-assisted reduction and maintenance

INTERVENTIONS:
Procedure: Percutaneous screw fixation through K-wire-assisted reduction and maintenance — Percutaneous screw fixation for acute scaphoid fractures through K-wire-assisted reduction and maintenance

SUMMARY:
The scaphoid is the most common fractured carpal bone in active adults, accounting for up to 80% of all carpal fractures. The optimum treatment approach of the acute scaphoid fractures is under discussion. Cast immobilization is the main treatment for non-displaced scaphoid fractures, however, about 20% of scaphoid fractures fail to heal with conservative treatment. Long periods of cast immobilization may result in wrist stiffness, loss of grip strength, muscle atrophy and disuse osteopenia. Operative treatment for displaced and unstable scaphoid fractures was mostly adopted, however, open fixation for scaphoid fractures have the inherent disadvantages of ligament and capsular dissection, blood vessels damage. This study introduces a novel measures of percutaneous screw fixation for acute scaphoid fractures. We used one K-wire maintaining the reduction of the scaphoid fractures throughout the entire process of drilling and screw insertion and screw fixation for acute scaphoid fractures.

ELIGIBILITY:
Inclusion Criteria:

* acute scaphoid fractures
* Injury to surgery less than 7 days
* Only one injured hand
* Written informed consent to undergo the surgical procedure
* Patients of either sex aged between 18 and 70 years

Exclusion Criteria:

* Patients with vascular injuried requiring revascularization
* Concomitant phalanx fractures or other injuries needing immobilization
* Loss of skin substance requiring grafts or flaps
* Uncompensated diabetes, neoplasia, haemocoagulative alterations, psychic disorders
* Smokers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
The modified Mayo wrist scoring system | 3 months
  The function outcomes including pain, work status, range of motion (Rom) and grip strength were assessed and graded as excellent, good , fair and poor.

CONTACTS AND LOCATIONS:
Overall Officials: Chunjie Liu, M.D., Study Chair — Hebei Medical University

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Yu Y, Cui H, Yang X, Yu X, Bai Y. A novel percutaneous achievement and maintenance of reduction and screw fixation for acute displaced scaphoid fractures: minimum two-year follow-up. Int Orthop. 2018 Aug;42(8):1911-1916. doi: 10.1007/s00264-018-3758-5. Epub 2018 Jan 10. PMID 29318360
- [Background] Merrell G, Slade J. Technique for percutaneous fixation of displaced and nondisplaced acute scaphoid fractures and select nonunions. J Hand Surg Am. 2008 Jul-Aug;33(6):966-73. doi: 10.1016/j.jhsa.2008.04.023. PMID 18656774
- [Background] Morsy M, Sabbagh MD, van Alphen NA, Laungani AT, Kadar A, Moran SL. The Vascular Anatomy of the Scaphoid: New Discoveries Using Micro-Computed Tomography Imaging. J Hand Surg Am. 2019 Nov;44(11):928-938. doi: 10.1016/j.jhsa.2019.08.001. Epub 2019 Sep 19. PMID 31543293
- [Background] Garcia RM, Ruch DS. Management of scaphoid fractures in the athlete: open and percutaneous fixation. Sports Med Arthrosc Rev. 2014 Mar;22(1):22-8. doi: 10.1097/JSA.0000000000000008. PMID 24651287